CLINICAL TRIAL: NCT02530281
Title: A Phase 3, Randomized, Double-Blind, Vehicle-Controlled Efficacy and Safety Study of Glycopyrronium in Subjects With Axillary Hyperhydrosis
Brief Title: Study of Glycopyrronium in Axillary Hyperhydrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Journey Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRM04-HH04; 2015-002052-27 (EudraCT Number)
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- glycopyrronium (Experimental): glycopyrronium Topical Wipes
  Interventions: Drug: glycopyrronium Topical Wipes
- Vehicle (Placebo Comparator): glycopyrronium Topical Wipes, Vehicle
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: glycopyrronium Topical Wipes — Topical wipes containing glycopyrronium
  Other Names: DRM04
  Arms: glycopyrronium
Other: Vehicle — Vehicle (placebo) topical wipes
  Arms: Vehicle

SUMMARY:
The study is a randomized, double-blind, vehicle controlled, parallel group study, designed to assess the efficacy and safety of glycopyrronium topical wipes, once daily, compared to vehicle in subjects with axillary hyperhidrosis.

DETAILED DESCRIPTION:
This is a randomized, double-blind vehicle controlled study to assess the efficacy and safety of glycopyrronium topical wipes compared to vehicle in subjects with axillary hyperhidrosis.

Safety will be assessed through lab tests, ECG, physical exams and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 9 years of age.
* Primary, axillary hyperhidrosis of at least 6 months duration
* Hyperhidrosis Disease Severity Scale (HDSS) of 3 or 4 at Baseline
* Axillary Sweating Daily Diary (ASDD) ≥ 4 at Baseline
* Sweat production of at least 50 mg over 5 minutes in each axilla assessed gravimetrically

Exclusion Criteria:

* Prior surgical procedure for hyperhidrosis.
* Prior axillary treatment with an anti-hyperhidrosis medical device (approved or investigational).
* Prior treatment with botulinum toxin (e.g., Botox®) for axillary hyperhidrosis within 1 year of Baseline/Day 1.
* Previous active treatment in the Dermira DRM04-HH01 or DRM04-HH02 clinical trials.
* Axillary use of nonprescription antiperspirants within 1 week or prescription antiperspirants within 2 weeks of Baseline.
* Subjects on new or regimens of psychotherapeutic medications that have changed within 2 months of baseline.
* Treatment with systemic anticholinergics within 4 weeks of the baseline visit unless dosing has been stable for at least 4 months.
* Other treatment with glycopyrrolate within 4 weeks prior to Baseline.
* Secondary axillary hyperhidrosis or presence of a condition that may cause secondary hyperhidrosis.
* History of Sjögren's syndrome or Sicca syndrome.
* History of glaucoma, inflammatory bowel disease, toxic megacolon, or febrile illness.
* Men with a history of urinary retention requiring catheterization due to prostatic hypertrophy or severe obstructive symptoms of prostatic hypertrophy.
* History or presence of ventricular arrhythmias, atrial fibrillation, atrial flutter.
* Other systemic diseases or active uncontrolled infections, or any other condition which, in the judgment of the Investigator, would put the subject at unacceptable risk for participation in the study.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne M Deans, MT, Study Director — Dermira, Inc.
Locations (31):
- United States (21):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Therapeutics Clinical Research, San Diego, California
  - Skin Care Research, Inc., Boca Raton, Florida
  - Study Protocol, Inc., Boynton Beach, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - Tory Sullivan, M.D., P.A., North Miami Beach, Florida
  - Research Institute of the Southeast, West Palm Beach, Florida
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Prairie Health and Wellness, Wichita, Kansas
  - St. Louis University Dermatology, St Louis, Missouri
  - Meridian Clinical Research, Omaha, Nebraska
  - Dermatology and Laser Center, Charleston, South Carolina
  - Rivergate Dermatology Clinical Research Center, PLLC, Goodlettsville, Tennessee
  - DermResearch, Austin, Texas
  - J&S Studies, College Station, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - ACRC Trials / Innovative Dermatology, Plano, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Charlottesville Dermatology Research Center, Charlottesville, Virginia
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Germany (10):
  - Klinik fur Dermatologie, Allergologie und Venerologie Allergie-Centrum-Charite, Berlin
  - Pro DERMA im Hautzentrum Dulmen, Dülmen
  - Medical Practice and Derma Study Center Friedrichshafen GmbH, Friedrichshafen
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Hautarztpraxis, Glückstadt
  - Tagesklinik DermaKiel, Kiel
  - Dermatolosche Gemeinschaftspraxis, Mahlow
  - Hautarztpraxis, Pinneberg
  - Gemeinschaftspraxis Weber & Cranic, Schweinfurt
  - Hautarztpraxis, Stuttgart

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hebert AA, Glaser DA, Green L, Hull C, Cather J, Drew J, Gopalan R, Pariser DM. Long-term efficacy and safety of topical glycopyrronium tosylate for the treatment of primary axillary hyperhidrosis: Post hoc pediatric subgroup analysis from a 44-week open-label extension study. Pediatr Dermatol. 2020 May;37(3):490-497. doi: 10.1111/pde.14135. Epub 2020 Mar 8. PMID 32147881
- [Derived] Glaser DA, Hebert AA, Nast A, Werschler WP, Green L, Mamelok RD, Quiring J, Drew J, Pariser DM. A 44-Week Open-Label Study Evaluating Safety and Efficacy of Topical Glycopyrronium Tosylate in Patients with Primary Axillary Hyperhidrosis. Am J Clin Dermatol. 2019 Aug;20(4):593-604. doi: 10.1007/s40257-019-00446-6. PMID 31111409
- [Derived] Pariser DM, Hebert AA, Drew J, Quiring J, Gopalan R, Glaser DA. Topical Glycopyrronium Tosylate for the Treatment of Primary Axillary Hyperhidrosis: Patient-Reported Outcomes from the ATMOS-1 and ATMOS-2 Phase III Randomized Controlled Trials. Am J Clin Dermatol. 2019 Feb;20(1):135-145. doi: 10.1007/s40257-018-0395-0. PMID 30378087

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glycopyrronium | Vehicle
Started | 229 | 115
Completed | 208 | 112
Not Completed | 21 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glycopyrronium | Vehicle | Total
Number analyzed (Participants) | 229 | 115 | 344
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 10 | 34
  Between 18 and 65 years | 204 | 101 | 305
  >=65 years | 1 | 4 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 60 | 190
  Male | 99 | 55 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 23 | 69
  Not Hispanic or Latino | 183 | 92 | 275
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 31 | 16 | 47
  White | 182 | 94 | 276
  More than one race | 10 | 3 | 13
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Have a ≥4-point Improvement in the Weekly Mean Score of ASDD Item #2 From Baseline at Week 4
Description: The Axillary Sweating Daily Diary (ASDD) is a 4-item instrument designed to measure the severity of axillary hyperhidrosis and its impact on daily activities. The 4 Items are:
  1. During the past 24 hours, did you have any underarm sweating? (Yes or No)
  2. During the past 24 hours, how would you rate your underarm sweating at its worst? (0=No sweating at all, 1, 2,…, 10=Worst possible sweating)
  3. During the past 24 hours, to what extent did your underarm sweating impact your activities? (0=Not at all, 1=A little bit, 2=A moderate amount, 3=A great deal and 4=An extreme amount)
  4. During the past 24 hours, how bothered were you by your underarm sweating? (0=Not at all bothered, 1=A little bothered, 2=Moderately bothered, 3=Very bothered, 4=Extremely bothered)
Time Frame: From Baseline to Week 4
Population: Participant
Measure: Number; unit: percent of subjects
Arm/Group | Glycopyrronium | Vehicle
Number analyzed (Participants) | 229 | 115
percent of subjects | 52.8 | 28.3
Statistical Analysis 1: Comparison: Glycopyrronium vs Vehicle; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel

2. Primary Outcome: Mean Absolute Change From Baseline in Gravimetrically-measured Sweat Production at Week 4
Description: Subjects are acclimated to the environment for 30 minutes. Dry gauze is weighed. The dry gauze is then applied to the subject's axilla with the arm down by the subject's side or on their lap during the 5-minute period of sweat production. The gauze with the sweat is then weighed. The difference between the Weight of the gauze with sweat and the dry gauze is the gravimetric sweat measurement in mg/5min.
Time Frame: From Baseline to Week 4
Population: Participant
Measure: Least Squares Mean (Standard Deviation); unit: mg/5 min
Arm/Group | Glycopyrronium | Vehicle
Number analyzed (Participants) | 229 | 115
mg/5 min | -102.00 (176.136) | -100.34 (172.276)
Statistical Analysis 1: Comparison: Glycopyrronium vs Vehicle; Test type: Other; p = 0.065, ANCOVA; Ranked ANCOVA

3. Primary Outcome: Median Absolute Change From Baseline in Gravimetrically-measured Sweat Production at Week 4
Time Frame: From Baseline to Week 4
Population: Participant
Measure: Median (Inter-Quartile Range); unit: mg/5 min
Arm/Group | Glycopyrronium | Vehicle
Number analyzed (Participants) | 229 | 115
mg/5 min | -80.79 [-148.78 to -40.15] | -65.81 [-105.67 to -27.65]
Statistical Analysis 1: Comparison: Glycopyrronium vs Vehicle; Test type: Other; p = 0.065, ANCOVA; Ranked ANCOVA

4. Primary Outcome: Mean Absolute Change From Baseline in Gravimetrically-measured Sweat Production at Week 4, Excluding Centers With Outlier Data
Time Frame: Baseline - Week 4
Population: Participant
Measure: Least Squares Mean (Standard Deviation); unit: mg/5 min
Arm/Group | Glycopyrronium | Vehicle
Number analyzed (Participants) | 220 | 110
mg/5 min | -100.56 (98.151) | -88.08 (95.695)
Statistical Analysis 1: Comparison: Glycopyrronium vs Vehicle; Test type: Other; p = 0.001, ANCOVA; Ranked ANCOVA

5. Secondary Outcome: Percentage of Subjects Who Have a ≥2 Grade Improvement in Hyperhidrosis Disease Severity Scale (HDSS) From Baseline at Week 4
Description: Hyperhidrosis Disease Severity Scale (HDSS) is a disease specific diagnostic tool that provides a qualitative measure of the severity of the subjects' condition based on how it affects daily activities.
  1 (Best), 2, 3, 4 (Worst)
Time Frame: From Baseline to Week 4
Population: Participant
Measure: Number; unit: percent of subjects
Arm/Group | Glycopyrronium | Vehicle
Number analyzed (Participants) | 229 | 115
percent of subjects | 56.5 | 23.7
Statistical Analysis 1: Comparison: Glycopyrronium vs Vehicle; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel

6. Secondary Outcome: Percentage of Subjects Who Have at Least a 50% Reduction in Gravimetrically Measured Sweat Production From Baseline at Week 4
Time Frame: From Baseline to Week 4
Population: Participant
Measure: Number; unit: percent of subjects
Arm/Group | Glycopyrronium | Vehicle
Number analyzed (Participants) | 229 | 115
percent of subjects | 72.4 | 53.2
Statistical Analysis 1: Comparison: Glycopyrronium vs Vehicle; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: up to 35 days
Description: The Total Participants at risk are based on the Safety population, defined as, Participants who were randomized and received at least one confirmed dose of study drug.
Arm/Group | Glycopyrronium | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/227 | 0/114
Serious Adverse Events (participants affected / at risk) | 1/227 | 0/114
Other Adverse Events (participants affected / at risk) | 68/227 | 16/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glycopyrronium (N=227) | Vehicle (N=114)
unilateral mydriasis (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Glycopyrronium (N=227) | Vehicle (N=114)
Dry Mouth (Gastrointestinal disorders) | 43 | 4
Application Site Pain (General disorders) | 20 | 11
Application Site Pruritis (General disorders) | 4 | 6
Mydriasis (Eye disorders) | 14 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes